CLINICAL TRIAL: NCT05760937
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single, Ascending Doses of BMS-986447 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability and Drug Levels of BMS-986447 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IM054-003
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Pharmacodynamics; Healthy Participants; BMS-986447

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986447 (Experimental)
  Interventions: Drug: BMS-986447
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986447 — Specified dose on specified days
  Arms: BMS-986447
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and drug levels of single, oral doses of BMS-986447 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kilograms per metered square (kg/m^2), inclusive.
* Healthy male and female participants without clinically significant deviation from normal in medical history, physical examination, ECG, and clinical laboratory determinations.
* A negative COVID-19 test, which will be performed in the manner mandated by the clinical side where the study is being conducted, at screening and check-in Day -2.

Exclusion Criteria:

* Participant has any condition that confounds the ability to interpret data from the study.
* Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if the participant was to participate in the study.
* Any major surgery or planned surgery (except gastrointestinal [GI] surgery, as described below) within 12 weeks of study intervention administration.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 59 days
Number of Participants with Serious AEs (SAEs) | Up to 59 days
Number of Participants with Clinical Laboratory Abnormalities | Up to 34 days
Number of Participants with Vital Sign Abnormalities | Up to 35 days
Number of Participants with Physical Examination Abnormalities | Up to 35 days
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to 34 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 72 hours postdose
Time of maximum observed plasma concentration (Tmax) | Up to 72 hours postdose
Apparent terminal phase half-life (T-Half) | Up to 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com